CLINICAL TRIAL: NCT00786968
Title: An Extension Study of Intrathecal Enzyme Replacement Therapy for Spinal Cord Compression in Mucopolysaccharidosis I
Brief Title: Extension Study of Intrathecal Enzyme Replacement Therapy for MPS I
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to slow enrolment.
Sponsor: Patricia I. Dickson, M.D. (Individual)
Collaborators: The Ryan Foundation (Other)
Responsible Party: Sponsor-Investigator, Patricia I. Dickson, M.D., Associate Professor of Pediatrics, Dickson, Patricia I., M.D.
Organization: Dickson, Patricia I., M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRC-001-01
Record Dates: First submitted 2008-06-17; First posted 2008-11-06 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Spinal Cord Compression; Mucopolysaccharidosis I; Hurler-Scheie Syndrome; Scheie Syndrome; Lysosomal Storage Disease
Keywords: mucopolysaccharidosis; Hurler-Scheie; Scheie; laronidase; spinal cord compression; central nervous system; enzyme replacement therapy; intrathecal
MeSH Terms: conditions — Spinal Cord Compression; Mucopolysaccharidosis I; Lysosomal Storage Diseases; Mucopolysaccharidoses | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intrathecal laronidase (Experimental): drug laronidase, dose 1.74 mg, route intrathecal, frequency every 30-90 days, duration 1 year
  Interventions: Drug: laronidase

INTERVENTIONS:
Drug: laronidase — 1.74 mg intrathecally every 1-3 months for 1 year
  Other Names: Aldurazyme; recombinant human alpha-l-iduronidase

SUMMARY:
This is a one-year extension study of the use of laronidase into the spinal fluid to treat spinal cord compression in mucopolysaccharidosis I. Mucopolysaccharidosis I is a rare genetic condition due to deficiency of the enzyme alpha-l-iduronidase. Spinal cord compression occurs in this condition due to accumulation of material called glycosaminoglycans (GAG). Laronidase is the manufactured form of the enzyme alpha-l-iduronidase that is deficient in mucopolysaccharidosis I patients. The aim of this study is to determine whether laronidase is safe and effective when given into the spinal fluid as a potential non-surgical treatment for spinal cord compression due to mucopolysaccharidosis I disease. Funding Source -- FDA OOPD

DETAILED DESCRIPTION:
Enzyme replacement therapy (ERT) has been developed for mucopolysaccharidosis I (MPS I), a lysosomal storage disorder. ERT helps many physical ailments due to the disease, but does not treat the central nervous system, due to inability to cross the blood brain barrier. Our purpose is to test delivery of ERT to the spinal fluid via intrathecal injection in patients with MPS I. In this pilot study, we will use recombinant human α-L-iduronidase administered intrathecally once per month for four months to individuals with the Hurler-Scheie and Scheie forms of MPS I and spinal cord compression. If successful, intrathecal delivery could represent a practical, straightforward method of treating central nervous system disease due to lysosomal storage.

ELIGIBILITY:
Inclusion Criteria:

* Hurler-Scheie, Scheie form of MPS I, or Hurler 2 years after hematopoietic stem cell transplantation

  * Spinal cord compression
  * Has received intrathecal laronidase previously with good response and no significant safety concerns
  * Age greater than 8 years
  * Able to provide legal informed consent
  * Aware of clinical treatment option of observation without treatment or surgical decompression
  * Negative urine pregnancy test at screening (nonsterile females of child-bearing potential who are sexually active only)

Exclusion Criteria:

* Severe (Hurler) form of MPS I
* Desires surgical or medical treatment of spinal cord compression
* Spinal cord compression that warrants immediate surgical intervention
* Pregnancy or lactation
* Hematopoietic stem cell transplantation within 2 years of study enrollment
* Receipt of an investigational drug within 30 days of enrollment
* Infusion reactions to laronidase that required medical intervention, prophylaxis, or altered enzyme administration
* Significant anti-iduronidase antibody titer
* Recent initiation of intravenous laronidase (within past 6 months)
* Presence of cervical subluxation or similar external pathology as the major cause of cord compression symptoms for which surgical intervention should be immediately undertaken

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
safety of intrathecal enzyme treatment by blood and spinal fluid tests; improvement or stabilization in neurologic signs and symptoms of spinal cord compression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Patricia I Dickson, MD, Principal Investigator — Los Angeles Biomedical Research Institute at Harbor-UCLA
Locations (2):
- Los Angeles Biomedical Research Institute at Harbor-UCLA, Torrance, California, United States
- Helsinki University Central Hospital, Helsinki, Finland